CLINICAL TRIAL: NCT03445169
Title: A Single-Dose, Open-Label, Randomized, Food Effect Study in Healthy Volunteers With PT2977 Tablets
Brief Title: A Food Effect Study in Healthy Volunteers With Belzutifan (PT2977, MK-6482) Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peloton Therapeutics, Inc., a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 6482-002; PT2977-103 (Other: Pelaton Study ID)
Record Dates: First submitted 2018-02-20; First posted 2018-02-26 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Healthy
MeSH Terms: interventions — belzutifan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fasting (Experimental): Belzutifan tablets taken after fasting
  Interventions: Drug: Belzutifan
- Non-Fasting (Experimental): Belzutifan taken after eating a high calorie meal
  Interventions: Drug: Belzutifan

INTERVENTIONS:
Drug: Belzutifan — Belzutifan Tablets
  Other Names: MK-6482,; PT2977

SUMMARY:
This Phase 1, single-dose study will be conducted in adult male and female subjects (N = 16) who are in general good health and selected for participation in the study according to the selection criteria. This study will assess the effect of food on the pharmacokinetics of belzutifan Tablets. The study will consist of two periods and will be conducted in a crossover fashion.

DETAILED DESCRIPTION:
Subjects will be randomized in equal numbers to two sequences of meal conditions (fasting and non-fasting). Serial blood samples will be collected after dose administration in each period. Subjects will be confined at the clinical research for a portion of each period.

ELIGIBILITY:
Inclusion Criteria:

* Female or vasectomized male;
* If of childbearing potential, willing to practice methods of birth control;
* If of childbearing potential, must be non-pregnant and non-lactating and have a negative serum pregnancy test result prior to enrollment into the trial;
* Has a body mass index (BMI) between 19 and 32 kg/m2; Willing and able to give written informed consent for study participation and provide consent for access to medical data;
* Willing and able to cooperate with all aspects of the protocol.

Exclusion Criteria:

* Any vaccination within 30 days before start of this study and throughout the study;
* Abnormal blood pressure or pulse rate;
* Abnormal screening electrocardiogram (ECG);
* Receipt of any investigational agent within 30 days;
* A positive history of drug abuse or a positive test result for drug(s) of abuse;
* Female subjects who are planning a pregnancy or are pregnant or lactating.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-02-23 (Actual); Primary Completion 2018-05-26 (Actual); Study Completion 2018-05-26 (Actual)

PRIMARY OUTCOMES:
Plasma Concentrations of belzutifan assessed in both the fasting and non-fasting conditions and compared | 9 days in each of the fasting and non-fasting arms
  Blood samples to assess concentrations of belzutifan will be collected throughout the sampling time frame

CONTACTS AND LOCATIONS:
Locations (1):
- Spaulding Clinical, West Bend, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php